CLINICAL TRIAL: NCT01033227
Title: A Safety and Efficacy Evaluation of Sodium Nitrite Injection for the Treatment of Vaso-Occlusive Crisis Associated With Sickle Cell Disease
Brief Title: Safety and Efficacy of Sodium Nitrite in Sickle Cell Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Hope Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Thomas Coates, Hematology Division Head, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SN-SC-02-01
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; sickle cell anemia; pain crisis; nitric oxide; nitrite; vaso occlusive crisis; pain medication; sickled cells; blood flow; microcirculation
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No drug (No Intervention): No study drug administered
- Sodium nitrite injection, USP (Experimental): Administration if sodium nitrite injection, USP
  Interventions: Drug: sodium nitrite injection, usp

INTERVENTIONS:
Drug: sodium nitrite injection, usp — Sodium nitrite injection, USP will be administered in blocks of six subjects (3 sodium nitrite and 3 no drug). A total of five dose levels are planned, pending safety starting. Drug will be given by continuous infusion infusion for 48 hours starting at 6 nmol/min/kg (10% of the maximal tolerated dose).
  Other Names: sodium nitrite
  Arms: Sodium nitrite injection, USP

SUMMARY:
This study will determine if administration of sodium nitrite is safe and can improve small vessel blood flow and tissue oxygenation when given as an additional treatment in patients with acute vaso-occlusive crisis (pain crisis) associated with sickle cell disease.

DETAILED DESCRIPTION:
Nitric oxide (NO) is a naturally occuring chemical that relaxes blood vessels and helps improve blood flow.

The pain associated with vaso-occlusive crisis (pain crisis) in sickle cell disease is caused in part by lack of oxygen and increased tissue acid because blood flow is blocked by stiff sickle red cells. Administration of sodium nitrite should generate nitric oxide in this area of hypoxia and acidosis and improve blood flow.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for admission to the study:

1. Male or female subject aged between 8 and 23 years of age; only patients up to the age of 23 will be studied at Childrens Hospital Los Angeles
2. Electrophoretic diagnosis of sickle cell disease;
3. Sudden onset of acute pain involving >=1 sites typical of vaso-occlusive crisis (Vaso-occlusive crisis is defined as acute, severe pain in the extremities, chest, abdomen, or back that can not be explained by other complications of sickle cell disease or by a cause other than sickle cell disease.);
4. Severe pain requiring parenteral analgesics and hospitalization.
5. Informed consent obtained from a legal representative or from subjects 18 years of age or older before enrollment;
6. Being willing and able to be followed for at least 30 days for evaluation.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Clinically significant bleeding;
2. Current drug abuse or participation in methadone program;
3. Episode of pain requiring hospitalization within 2 weeks prior to current admission;
4. Other complications of sickle cell disease including cerebrovascular accident, pulmonary hypertension, or seizure;
5. Pregnancy (confirmed by a serum human chorionic gonadotropin pregnancy test) or breast feeding;
6. Blood pressure less than 25th percentile for the subject's age and sex on admission or at the time of screening;
7. Methemoglobinemia >3%;
8. Anemia with hemoglobin level less than 6 g/dL;
9. Red blood cell G6PD deficiency, by laboratory testing prior to enrollment;
10. History of allergy to nitrites or allergy to other substances characterized by dyspnea and cyanosis;
11. Treatment with allopurinol, a medication that could interfere with nitrite metabolism, within the past 30 days before screening;
12. Treatment with any investigational drug within the past 30 days;
13. Significant acute or chronic concomitant diseases (including renal, hepatic, cardiovascular, pulmonary, or oncologic disease, sepsis, pulmonary edema, pulmonary embolism) that would be inconsistent with survival for at least 6 months;
14. Any subject judged by the clinical investigator or study manager to be inappropriate for the study.

Ages: 8 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Coates, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood KC, Hsu LL, Gladwin MT. Sickle cell disease vasculopathy: a state of nitric oxide resistance. Free Radic Biol Med. 2008 Apr 15;44(8):1506-28. doi: 10.1016/j.freeradbiomed.2008.01.008. Epub 2008 Jan 26. PMID 18261470
- [Background] Mack AK, McGowan Ii VR, Tremonti CK, Ackah D, Barnett C, Machado RF, Gladwin MT, Kato GJ. Sodium nitrite promotes regional blood flow in patients with sickle cell disease: a phase I/II study. Br J Haematol. 2008 Sep;142(6):971-8. doi: 10.1111/j.1365-2141.2008.07259.x. Epub 2008 Jul 11. PMID 18671702
- [Background] Lundberg JO, Weitzberg E. Nitrite reduction to nitric oxide in the vasculature. Am J Physiol Heart Circ Physiol. 2008 Aug;295(2):H477-8. doi: 10.1152/ajpheart.00611.2008. Epub 2008 Jun 27. No abstract available. PMID 18586886
- [Background] Hachiya T, Blaber AP, Saito M. Near-infrared spectroscopy provides an index of blood flow and vasoconstriction in calf skeletal muscle during lower body negative pressure. Acta Physiol (Oxf). 2008 Jun;193(2):117-27. doi: 10.1111/j.1748-1716.2007.01827.x. Epub 2007 Dec 19. PMID 18162057
- [Background] Cappellini MD, Fiorelli G. Glucose-6-phosphate dehydrogenase deficiency. Lancet. 2008 Jan 5;371(9606):64-74. doi: 10.1016/S0140-6736(08)60073-2. PMID 18177777
- [Background] Villagra J, Shiva S, Hunter LA, Machado RF, Gladwin MT, Kato GJ. Platelet activation in patients with sickle disease, hemolysis-associated pulmonary hypertension, and nitric oxide scavenging by cell-free hemoglobin. Blood. 2007 Sep 15;110(6):2166-72. doi: 10.1182/blood-2006-12-061697. Epub 2007 May 29. PMID 17536019
- [Background] Vanin AF, Bevers LM, Slama-Schwok A, van Faassen EE. Nitric oxide synthase reduces nitrite to NO under anoxia. Cell Mol Life Sci. 2007 Jan;64(1):96-103. doi: 10.1007/s00018-006-6374-2. PMID 17160351
- [Background] Kato GJ, McGowan V, Machado RF, Little JA, Taylor J 6th, Morris CR, Nichols JS, Wang X, Poljakovic M, Morris SM Jr, Gladwin MT. Lactate dehydrogenase as a biomarker of hemolysis-associated nitric oxide resistance, priapism, leg ulceration, pulmonary hypertension, and death in patients with sickle cell disease. Blood. 2006 Mar 15;107(6):2279-85. doi: 10.1182/blood-2005-06-2373. Epub 2005 Nov 15. PMID 16291595
- [Background] Ferreira LF, Harper AJ, Townsend DK, Lutjemeier BJ, Barstow TJ. Kinetics of estimated human muscle capillary blood flow during recovery from exercise. Exp Physiol. 2005 Sep;90(5):715-26. doi: 10.1113/expphysiol.2005.030189. Epub 2005 May 20. PMID 15908509
- [Background] Raj A, Bertolone SJ, Mangold S, Edmonds HL Jr. Assessment of cerebral tissue oxygenation in patients with sickle cell disease: effect of transfusion therapy. J Pediatr Hematol Oncol. 2004 May;26(5):279-83. doi: 10.1097/00043426-200405000-00004. PMID 15111778
- [Background] Gladwin MT, Crawford JH, Patel RP. The biochemistry of nitric oxide, nitrite, and hemoglobin: role in blood flow regulation. Free Radic Biol Med. 2004 Mar 15;36(6):707-17. doi: 10.1016/j.freeradbiomed.2003.11.032. PMID 14990351
- [Background] Gladwin MT, Lancaster JR Jr, Freeman BA, Schechter AN. Nitric oxide's reactions with hemoglobin: a view through the SNO-storm. Nat Med. 2003 May;9(5):496-500. doi: 10.1038/nm0503-496. No abstract available. PMID 12724752
- [Background] Cosby K, Partovi KS, Crawford JH, Patel RP, Reiter CD, Martyr S, Yang BK, Waclawiw MA, Zalos G, Xu X, Huang KT, Shields H, Kim-Shapiro DB, Schechter AN, Cannon RO 3rd, Gladwin MT. Nitrite reduction to nitric oxide by deoxyhemoglobin vasodilates the human circulation. Nat Med. 2003 Dec;9(12):1498-505. doi: 10.1038/nm954. Epub 2003 Nov 2. PMID 14595407
- [Background] Gladwin MT, Schechter AN, Shelhamer JH, Ognibene FP. The acute chest syndrome in sickle cell disease. Possible role of nitric oxide in its pathophysiology and treatment. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1368-76. doi: 10.1164/ajrccm.159.5.9810094. No abstract available. PMID 10228097
- [Background] Lundberg JO, Gladwin MT, Ahluwalia A, Benjamin N, Bryan NS, Butler A, Cabrales P, Fago A, Feelisch M, Ford PC, Freeman BA, Frenneaux M, Friedman J, Kelm M, Kevil CG, Kim-Shapiro DB, Kozlov AV, Lancaster JR Jr, Lefer DJ, McColl K, McCurry K, Patel RP, Petersson J, Rassaf T, Reutov VP, Richter-Addo GB, Schechter A, Shiva S, Tsuchiya K, van Faassen EE, Webb AJ, Zuckerbraun BS, Zweier JL, Weitzberg E. Nitrate and nitrite in biology, nutrition and therapeutics. Nat Chem Biol. 2009 Dec;5(12):865-9. doi: 10.1038/nchembio.260. PMID 19915529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for the study during regular clinic visits.
Pre-assignment Details: Once consent signed subjects would not be randomized into the treatment arm until (if or when) they had their admission to the hospital for vaso-occlusive crisis (VOC).
Groups:
- No Drug: This group did not receive anything additional in the no drug arm. The treatment group received the study drug and the non treatment group received no drug.
Period: Overall Study
Arm/Group | No Drug | Sodium Nitrite Injection, USP
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Drug | Sodium Nitrite Injection, USP | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 16 [15 to 17] | 15.5 [11 to 20] | 16 [11 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Sickle Cell Disease hb SS [Count of Participants; unit: Participants] | 3 | 1 | 4
Sbeta+thalassemia [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 48 Hour Sodium Nitrite Infusion Safety as Determined by Number of Participants With No Adverse Events
Description: The primary end points will be to determine if a) a 48-hour sodium nitrite infusion is tolerated without a decrease in mean arterial blood pressure by 15mmHg for greater than 2 hours or development of methemoglobin greater than 5% and b) a 48-hour sodium nitrite infusion is safe as determined by monitoring for adverse events
Time Frame: 48 hours from start of infusion
Measure: Count of Participants; unit: Participants
Groups:
- No Drug: Will not receive study drug, there is no placebo in this study. The patient will know they are not receiving the study drug.
- Sodium Nitrite Injection, USP: Administration of sodium nitrite injection, USP
Arm/Group | No Drug | Sodium Nitrite Injection, USP
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

2. Secondary Outcome: Secondary End Point
Description: a) reduced the duration and intensity of pain; b) reduced total narcotic analgesic consumption; and c) reduced length of hospitalization.
Time Frame: 48 hours
Population: Data were *not collected* and the Outcome was never analyzed, study terminated
Arm/Group | No Drug | Sodium Nitrite Injection, USP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after completion of study drug
Groups:
- No Drug: This group received no study drug and no placebo. They received standard of care treatment.
Arm/Group | No Drug | Sodium Nitrite Injection, USP
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes